CLINICAL TRIAL: NCT04510896
Title: InheRET: A Software-as-a-Service (SaaS) Solution to Identifying Patients at Increased Risk for Hereditary Disease
Brief Title: Inherited Risk Evaluation Tool (InheRET): Identifying Patients at Increased Risk for Hereditary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: InheRET, Inc (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R41CA239842-01 (NIH)
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hereditary Cancer-Predisposing Syndrome
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Intervention Model Description: Each patient is requested to take the InheRET personal and family health history form. If consented patients fail to complete the form within one week of consenting, they may receive up to three (3) weekly reminder emails. The survey will take less than 10 minutes for low-risk patients. Completion time for higher risk patients depends on the size of the family, the number of conditions to report, and the patient's skill level with completing online forms. The InheRET form can be completed from any web-enabled device at the patient's convenience. Follow-up surveys will be sent as follows:
  1. Consented participants fail to complete the InheRET health history for 2 months after consent to determine reason(s) for not completing.
  2. Consented participants who complete the InheRET health history - 6 and 12 months after completion to identify actions taken since completion including genetic counseling, genetic testing, screening, lifestyle changes, and prophylaxis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-InheRET (No Intervention): Determine appropriate genetic counseling referral rates (as defined by NCCN guidelines) per patient (across all sites) in the pre-intervention 6-month period. Only referrals to Michigan Medicine (MM) genetics clinics will be included in the statistical analysis. Having access to MM health records, we will be able to assess the appropriateness of the referrals.
- Post-InheRET (Experimental): Determine appropriate genetic counseling referral rates (as defined by NCCN guidelines) per patient (across all sites) in the post-intervention period. Only referrals to Michigan Medicine genetics clinics will be included in the statistical analysis. Having access to MM health records, we will be able to assess the appropriateness of the referrals.
  Interventions: Other: InheRET; Other: Patient Acceptance; Other: Physician Acceptance Survey

INTERVENTIONS:
Other: InheRET — Primary Appropriate Referral Rates 6-months pre-intervention vs post-intervention Compare appropriate genetic counseling referral rates (as defined by NCCN guidelines) per patient (across all sites) in the pre-intervention vs post- intervention period. Only referrals to Michigan Medicine genetics clinics will be included in the statistical analysis. Having access to MM health records, we will be able to assess the appropriateness of the referrals.
  Other Names: InheRET 2.0 - Phase I; InheRET 3.0 - Phase II
  Arms: Post-InheRET
Other: Patient Acceptance — Acceptance by Patients Over the course of the study Acceptance measures will include completion rates and levels of ease of use of InheRET by the patient. Impact measures will include uptake of advised risk management interventions. We will qualitatively describe why patients do not follow up with their referral. We will explore patterns of acceptance and impact levels by demographic and clinical data using correlation, t- tests, ANOVA, or their non-parametric equivalents.
  Arms: Post-InheRET
Other: Physician Acceptance Survey — Secondary Acceptance by Physicians Over the course of the study Acceptance by physicians will measure the physician effort required to deploy and use InheRET in their respective clinics, and overall satisfaction. Impact measures will include appropriate referral rates and rates of genetic testing. We will qualitatively describe why patients are not referred for genetic counseling if indicated. We will explore patterns in acceptance and impact levels by demographic and clinical data using correlations, t-tests, ANOVA, or their non-parametric equivalents.
  Arms: Post-InheRET

SUMMARY:
This study will evaluate the impact InheRET™, an online family history gathering and risk assessment reporting tool, has on facilitating National Comprehensive Cancer Network(NCCN) guideline compliant referrals for cancer genetic counseling/genetic evaluation by decreasing and/or removing the barriers of 1) time-consuming in-clinic 3-generation family history collection, and 2) interpretation of the family and personal history in light of current NCCN guidelines.

Identifying individuals at increased risk for cancer has been shown to decrease morbidity and mortality in multiple clinical settings. Investigators hypothesize that InheRET will prove to be accurate, efficient, and accessible, and that its use will improve identification of individuals at risk for inherited susceptibility to cancer. The investigators propose also that using this tool will result in a reduction of inappropriate genetic counseling referrals and reduce unnecessary genetic testing in both primary and specialty care settings. InheRET will allow health care providers to focus resources on individuals at higher risk for developing cancer.

DETAILED DESCRIPTION:
This study will evaluate the impact InheRET™, an online family history gathering and risk assessment reporting tool, has on facilitating National Comprehensive Cancer Network(NCCN) guideline compliant referrals for cancer genetic counseling/genetic evaluation by decreasing and/or removing the barriers of 1) time-consuming in-clinic 3-generation family history collection, and 2) interpretation of the family and personal history in light of current NCCN guidelines.

This is a prospective study with a pre/post intervention analysis. The prior 6-months' genetic counseling referrals to Michigan Medicine will be collected for each site to serve as baseline data and compared to the intervention data to measure the difference made by InheRET utilization. Primary care sites are selected to offer the broadest range of patient populations to ensure the InheRET tool works well in diverse groups accessing varied clinical settings. The Cancer Genetics and MM Breast and Ovarian Cancer Risk Evaluation Clinics will allow us to measure the appropriateness of referrals and the impact of InheRET on genetic counseling workflows as patients from the primary care sites are referred for counseling from throughout the tri-state catchment areas and beyond. Similarly, investigators will review electronic health records for appropriateness of referrals to other counseling clinics at Michigan Medicine.

This will be accomplished by implementing InheRET in a variety of clinical settings to measure its acceptance by providers and patients as well as any changes made in referral patterns as a result of its use, compared to patterns of referral before it is implemented. Patients completing the InheRET online tool form will be followed longitudinally by surveys to discover their risk management actions (i.e. genetic counseling appointment, genetic testing, screenings, prophylaxis) and the reasons for or against undertaking such actions. Providers will also be surveyed to determine the impact InheRET has made to their workflow, the acceptability of this tool by their practice, and the usefulness of InheRET's features to accomplish its goals. This study has a goal enrollment of 2109 patients in Phase I (already enrolled) and at least 1023 patient subjects in Phase II (anticipated) to use the InheRET program for the purpose of this study and will also enroll six to twelve (6-12) physicians to obtain reflection on experience using InheRET for the purpose of this study.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care sites:Adult patients with New and Health Maintenance Exam appointments at participating clinics
* Genetics sites: Adult patients with new referrals for genetic counseling

Exclusion Criteria:

* Patients who were previously referred or who have an appointment for genetic counseling pending.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2232 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Pre- and Post-Rate of Referrals of Patients to Genetic Counseling from Primary Care Clinics, | 6 months prior to InheRET as compared to post implementation.
  Average number of patients per month referred to genetic counseling before and after InheRET's implementation in clinic.

SECONDARY OUTCOMES:
Physician Acceptance and Impact | Physicians will be surveyed within 3 months and again upon completion of enrollment, approximately 1 year.
  Physicians will be consented and surveyed to determine acceptance, utility, and impact on clinical workflows. For discrete data elements, data will be reported as the number of physicians out of "n" responses. Qualitative data will be anonymized as needed, grouped thematically and reported. Responses from the two surveys will be compared to determine if perceptions have changed over time. Data will be reported as above with a % change added for discrete data elements.
Patient Acceptance of InheRET | Immediately upon completion of the personal and family health history form.
  Acceptance measures will include InheRET program completion rates (%) and levels of ease of use of InheRET by the patient, via survey at completion of the form. Patients will rank, using a 5-point Likert Scale, Ease of Use, and Understandability. Yes/No answers with comments will collect data on Cancer Coverage, Increased Knowledge of Family History, and Problems Encountered.
  Investigators will explore patterns of acceptance levels by demographic and clinical data using correlation, t- tests, ANOVA, or their non-parametric equivalents.
Qualitative Impact on Patients | Follow up surveys 12- to 18-months following completion of the InheRET program.
  Impact measures will include uptake of advised risk management interventions (genetic counseling, testing, screening, lifestyle changes, therapeutics, and prophylaxis), collected by survey and through medical record exam. Investigators will also qualitatively describe why patients do not follow up with their referral, gathered through a survey sent 12 months after completion (Phase I) and every 6 months x 3 (Phase II). We will explore patterns of impact levels by demographic and clinical data using correlation, t- tests, ANOVA, or their non-parametric equivalents.

CONTACTS AND LOCATIONS:
Overall Officials: David Keren, MD, Principal Investigator — InheRET, Inc; Elena Stoffel, MD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - InheRET, Inc., Ann Arbor, Michigan
  - Michigan Medicine, Ann Arbor, Michigan
  - Hamilton Community Health Network - withdrew from study, Flint, Michigan
  - Ascension St. Mary's Hospital - withdrew from study, Saginaw, Michigan

IPD SHARING:
Plan to Share IPD: No
At this time, we do not plan to make individual participant data available for other researchers. Consolidated data will be available.